CLINICAL TRIAL: NCT00528437
Title: NYU 05-40 PBMTC ONC-032P:High Dose Temozolomide,Thiotepa and Carboplatin With Autologous Stem Cell Rescue (ASCR) Followed by Continuation Therapy With 13-cis-retinoic Acid in Patients With Recurrent/Refractory Malignant Brain Tumors
Brief Title: Temozolomide,Thiotepa and Carboplatin With Autologous Stem Cell Rescue Followed by 13-cis-retinoic Acid in Patients With Recurrent/Refractory Malignant Brain Tumors
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: NYU Langone Health (Other)
Collaborators: Children's Hospitals and Clinics of Minnesota (Other); Schneider Children's Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 12853; PBMTC ONC-032P (Other: Pediatric Blood and Marrow Tranplant Consortium)
Record Dates: First submitted 2007-09-10; First posted 2007-09-12 (Estimated); Results first posted 2021-07-08 (Actual); Last update posted 2021-07-08 (Actual); Status verified 2021-06

CONDITIONS: Brain Tumors
Keywords: Recurrent or refractory medulloblastoma/PNET; CNS germ cell tumors; Ependymomas; AT/RT; High grade glioma; Other malignant brain tumors
MeSH Terms: conditions — Brain Neoplasms; Recurrence; Ependymoma; Glioma | interventions — Temozolomide; Thiotepa; Carboplatin; Isotretinoin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Myeloablative Chemo-Temozolomide, Thiotepa, and Carboplatin. (Other)
  Interventions: Drug: temozolomide, thiotepa, carboplatin, 13-cis-retinoic acid

INTERVENTIONS:
Drug: temozolomide, thiotepa, carboplatin, 13-cis-retinoic acid — 13-cis-retinoic acid, when absorbed, may be subject to first-pass metabolism and subsequent plasma (and tumor) concentrations will depend on the rate of metabolism to the inactive 4-oxo metabolite.

SUMMARY:
The purpose of this study is to:

Find out how safe and effective (by monitoring the good and/or bad effects) treatment with high dose temozolomide, thiotepa and carboplatin with stem cell rescue followed by 13-cis-retinoic acid has on children and adolescents with recurrent/refractory brain tumors

Find out how the body uses 13-cis-retinoic acid by studying the your blood levels and proteins in the blood that break down the 13-cis-retinoic acid

Determine how well 13-cis-retinoic acid penetrates into the spinal fluid.

DETAILED DESCRIPTION:
Researchers have used high doses of combination chemotherapy followed by a stem cell rescue to treat recurrent brain tumors with moderate success. High dose chemotherapy with stem cell rescue has resulted in long term survival of about 25% in patients with several different types of recurrent brain tumors. Stem cells are cells in the bone marrow that produce blood cells. The stem cells are collected from the blood of the patient before the high dose chemotherapy. Patients are given high doses of chemotherapy to kill every brain tumor cell, but in the process the cells of the bone marrow are also killed. The previously collected stem cells are then infused into the patient to rescue the bone marrow and allow for healthy blood cells to re-populate and grow in the bone marrow. Initial studies used the drug etoposide along with carboplatin and thiotepa for the high dose chemotherapy. Patients had severe side effects, especially severe mouth-sores, thought mainly due to the etoposide, and some patients died from these side effects.

Recent studies have shown that a new drug, temozolomide, is active against some types of brain tumors. When it was given as a single drug to children with solid tumors, the side effects were considered to be tolerable. Temozolomide is given by mouth. In this study, researchers want to give high dose chemotherapy that includes the drugs temozolomide in place of etoposide, along with thiotepa and carboplatin. Patients will then be given their own stem cells back to rescue the bone marrow from the chemotherapy. A preliminary trial using this new drug combination was performed and has shown that patients tolerate this drug combination, even at the very high doses that will be used in this protocol.

Another drug that is being used in pediatric cancer treatment is called 13-cis-retinoic acid. This drug is closely related to vitamin A. It is taken by mouth. Cancer cells are immature cells that have not "grown up" into adult cells that do work in the body. 13-cis-retinoic acid is thought to act on some types of cancer cells to make them mature into cells that function in the body. It has also been shown in the laboratory to cause some brain tumor cells to undergo apoptosis. It has been used in other types of pediatric cancers and research is just beginning to use it for treatment of recurrent brain tumors. In this study researchers want to give you 13-cis-retinoic acid for 6 months after you recover from the high dose chemotherapy with stem cell rescue.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with recurrent or refractory medulloblastoma/PNET, CNS germ cell tumors, ependymomas, AT/RT, high grade glioma and other malignant brain tumors. Brainstem gliomas are eligible if residual disease is < 1.5cc and if the patient is off decadron.
2. Patients must have recurrent or refractory disease following at least one prior course of therapy and must have minimal residual disease defined as < 1.5 cm2 of enhancement. Patients with + CSF cytology, linear or fine nodular leptomeningeal disease are eligible.
3. Adequate hematologic, renal, liver, and cardiac function as demonstrated by laboratory values performed within 21 days, inclusive, prior to administration of temozolomide.
4. Patients must have an adequate number of autologous stem cells available defined as a minimum of 2 x 106 CD 34+ cells/kg and preferably at least 5 x 106 CD 34+ cells/kg.

Exclusion Criteria:

1. Previous myeloablative therapy
2. Frequent vomiting or medical condition that could interfere with oral medication intake (e.g., partial bowel obstruction)
3. Previous or concurrent malignancies at other sites with the exception of surgically cured carcinoma in-situ of the cervix and basal or squamous cell carcinoma of the skin. Patients with prior malignancies which have not required anti-tumor treatment within the preceding 24 months are eligible.

Ages: 6 Months to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 46 (Actual)
Dates: Start 2005-10 (Actual); Primary Completion 2017-06-30 (Actual); Study Completion 2017-12-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sharon L Gardner, MD, Principal Investigator — NYU Langone Health
Locations (17):
- United States (16):
  - Phoenix Children's Hospital, Phoenix, Arizona
  - Emory University, Atlanta, Georgia
  - Hawaii Pacific Health, Lihue, Hawaii
  - Children's Memorial Hospital, Chicago, Illinois
  - Riley Hospital for Children, Indianapolis, Indiana
  - Children's Hospital and Clinics of Minnesota, Minneapolis, Minnesota
  - Roswell Park Cancer Institute, Buffalo, New York
  - Steven and Alexandra Cohen Children's Medical Center of New York- North Shore LIJ, New Hyde Park, New York
  - NYU Hassenfeld Center, New York, New York
  - Nationwide Children's Hospital, Columbus, Ohio
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Medical Univ. of South Carolina, Charleston, South Carolina
  - Vanderbilt Univ., Nashville, Tennessee
  - Children's Medical Center of Dallas, Dallas, Texas
  - MD Anderson Cancer Center (MDACC), Houston, Texas
  - Virginia Commonwealth Univ., Richmond, Virginia
- Princess Margaret Hospital, Toronto, Ontario, Canada

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Myeloablative Chemo-Temozolomide, Thiotepa, and Carboplatin.
Started | 46
Completed | 46
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Myeloablative Chemo-Temozolomide, Thiotepa, and Carboplatin.
Number analyzed (Participants) | 46
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 40
  Between 18 and 65 years | 6
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15
  Male | 31
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 7
  Not Hispanic or Latino | 39
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 25
  More than one race | 0
  Unknown or Not Reported | 19
Region of Enrollment [Number; unit: participants]
  United States | 46

OUTCOME MEASURES:

1. Primary Outcome: Event-free Survival (EFS)
Description: EFS will be reported in patients with recurrent or refractory medulloblastoma/ primitive neuroectodermal tumors. EFS is defined as the length of time after primary treatment for a cancer ends that the patient remains free of certain complications or events that the treatment was intended to prevent or delay.
Time Frame: Day +42
Population: Efforts were made to contact the PI/study team members, but were unsuccessful. No study data are available
Arm/Group | Myeloablative Chemo-Temozolomide, Thiotepa, and Carboplatin.
Number analyzed (Participants) | 0

2. Primary Outcome: Overall Survival (OS)
Description: OS will be reported in patients with recurrent or refractory medulloblastoma/ primitive neuroectodermal tumors. OS is defined as the length of time from the start of treatment that patients diagnosed with disease are still alive.
Time Frame: Day +77
Population: Efforts were made to contact the PI/study team members, but were unsuccessful. No study data are available
Arm/Group | Myeloablative Chemo-Temozolomide, Thiotepa, and Carboplatin.
Number analyzed (Participants) | 0

3. Secondary Outcome: Toxicity of of 13-cis-retinoic Acid
Description: To report the toxicity of of 13-cis-retinoic acid following high dose temozolomide, thiotepa and carboplatin with ASCR.
Time Frame: One year
Population: Efforts were made to contact the PI/study team members, but were unsuccessful. No study data are available
Arm/Group | Myeloablative Chemo-Temozolomide, Thiotepa, and Carboplatin.
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Efforts were made to contact the PI/study team members, but were unsuccessful. No study data are available.
Description: Efforts were made to contact the PI/study team members, but were unsuccessful. No study data are available
Arm/Group | Myeloablative Chemo-Temozolomide, Thiotepa, and Carboplatin.
All-Cause Mortality (participants affected / at risk) | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2011-02-18): https://cdn.clinicaltrials.gov/large-docs/37/NCT00528437/Prot_SAP_ICF_000.pdf